CLINICAL TRIAL: NCT02478190
Title: ED Management of Severe Hyperglycemia: An Open-Label Randomized Clinical Trial
Brief Title: ED Management of Severe Hyperglycemia: A Clinical Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hennepin Healthcare Research Institute (Other)
Responsible Party: Principal Investigator, Brian Driver, Principal Investigator, Hennepin Healthcare Research Institute
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 15-3931
Record Dates: First submitted 2015-06-17; First posted 2015-06-23 (Estimated); Last update posted 2018-03-21 (Actual); Status verified 2018-03

CONDITIONS: Hyperglycemia; Diabetes Mellitus; Complications of Diabetes Mellitus; Diabetes-Related Complications; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Hyperglycemia; Diabetes Mellitus; Diabetes Complications; Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Tight control (Experimental): Patients in this arm will have a treatment glucose value at ED discharge of 350 mg/dL or lower.
  Interventions: Other: Tight control: goal glucose 350 mg/dL or lower
- Loose control (Experimental): Patients in this arm will have a treatment glucose value at ED discharge of 600 mg/dL or lower.
  Interventions: Other: Loose control: goal glucose 600 mg/dL or lower

INTERVENTIONS:
Other: Tight control: goal glucose 350 mg/dL or lower — Goal glucose at discharge will be 350 mg/dL or less.
  Arms: Tight control
Other: Loose control: goal glucose 600 mg/dL or lower — Goal glucose at discharge will be 600 mg/dL or less.
  Arms: Loose control

SUMMARY:
Emergency Department (ED) patients with severe hyperglycemia will be randomized to two treatment goals: discharge glucose less than 600 mg/dL or less than 350 mg/dL.

Randomization is stratified by whether the chief complaint is "High Blood Sugar" in the electronic medical record or other.

DETAILED DESCRIPTION:
It is common practice to provide insulin and/or intravenous (IV) fluids to lower glucose levels prior to discharge in patients that present with hyperglycemia. There is, however, no data supporting this practice.

A recent retrospective observational cohort study (HSR# 12-3497) of 567 ED patients with severe hyperglycemia demonstrated no association between discharge glucose levels and short-term adverse outcomes at 7 days (return ED visits, diabetic ketoacidosis (DKA), hospitalization, and death).

There were no other short-term adverse outcomes associated with the degree of glycemic control. Less than 1% of patients developed DKA at 7 days. No patients died.

As this was a retrospective study, the conclusions that can be drawn are limited by the lack of randomization and control; it is necessary to conduct a randomized controlled trial to quantify how much time is expended caring for these patients, and gather safety data.

This is important because much time and money is focused on glucose reduction, which may not change short-term outcomes. Furthermore, in retrospective analysis approximately 1.5% of patients receiving therapy for hyperglycemia developed iatrogenic hypoglycemia during the ED stay.

To detect a difference in length of stay by 60 minutes (Standard deviation is 100 minutes) with an p=0.05 and b=0.8, enrollment of 45 patients per group will be required, with a total enrollment of 90 patients. Enrollment will stop when 45 patients in each group have been contacted in follow-up.

This study will only include patients who are discharged from the ED. Patients who are enrolled and then eventually admitted to the hospital will be tabulated but excluded from the length of stay analysis.

Statistical analysis will be completed for the primary outcome with a Mann-Whitney U test, assuming the data will not be normally distributed. Secondary outcomes will be compared with chi-squared testing. A secondary regression model will be formed, based on covariates that could influence ED length of stay, such as amount of diagnostic testing completed.

ELIGIBILITY:
Inclusion Criteria:

* Glucose of more than 400mg/dL but less than 600 mg/dL at any point in the ED
* Working phone number and willing to discuss health status at 7-10 days via phone

Exclusion Criteria:

* Plan for hospital admission
* Already received insulin during the ED stay
* Type 1 diabetes
* Less than 18 years old
* Non-English speaking
* Altered mental status or encephalopathy (unable to provide informed consent)
* DKA, as determined clinically by the treating physician, without a lab requirement.
* Critically ill, as determined by the treating physician.
* Unable to provide informed consent
* Prisoners
* Pregnant women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2015-06 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
ED Length of Stay | This outcome measure is defined as the amount of time elapsed between when the patient is roomed, and when a discharge order is placed, during a single ED encounter, which is generally less than 4 hours.
  Time elapsed from when the patient is roomed until the time the MD places discharge order, by review of the Electronic Medical record by a blinded abstractor.

SECONDARY OUTCOMES:
Iatrogenic hypoglycemia | The patient will be followed during a single ED encounter, which is generally less than 4 hours.
  Rate of iatrogenic hypoglycemia in both groups, defined as: glucose <60 or glucose less than 100 mg/dL and symptoms of hypoglycemia that resolved with food/drink, or any use of IV dextrose 50%, glucagon, or oral glucose tabs/gel
Return ED visit for hyperglycemia and hospital admission for any reason, excluding trauma | 7 days
  Composite outcome of rate of repeat ED visit for hyperglycemia or hospital admission for any reason, excluding trauma admission. ED visit for hyperglycemia defined as: chief complaint of hyperglycemia, chief complaint of polyuria, polydipsia, fatigue, blurry vision, or malaise and found to have blood glucose more than 250 mg/dL, primary ED diagnosis of hyperglycemia, or ED or hospital diagnosis of DKA or hyperosmolar syndrome.
Return ED visit for any reason | 7 days
  Each patient will be assessed via chart review and telephone follow up to see if they visited an ED for any reason during the 7 day time frame. Rates of ED visits for any reason at 7 days will be compared between the two treatment arms.

CONTACTS AND LOCATIONS:
Overall Officials: Brian Driver, MD, Principal Investigator — HCMC
Locations (1):
- Hennepin County Medical Center, Minneapolis, Minnesota, United States

REFERENCES:
- [Derived] Driver BE, Klein LR, Cole JB, Prekker ME, Fagerstrom ET, Miner JR. Comparison of two glycemic discharge goals in ED patients with hyperglycemia, a randomized trial. Am J Emerg Med. 2019 Jul;37(7):1295-1300. doi: 10.1016/j.ajem.2018.09.053. Epub 2018 Oct 5. PMID 30316635